CLINICAL TRIAL: NCT05201495
Title: A Clinical Evaluation of the Jewel P-WCD in Subjects at High Risk for Sudden Cardiac Arrest
Brief Title: The Jewel IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Element Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-2053
Record Dates: First submitted 2022-01-05; First posted 2022-01-21 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Sudden Cardiac Arrest
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Jewel Patch Wearable Cardioverter Defibrillator (P-WCD)
  Interventions: Device: Jewel Patch Wearable Cardioverter Defibrillator (P-WCD)

INTERVENTIONS:
Device: Jewel Patch Wearable Cardioverter Defibrillator (P-WCD) — Automatic external cardioverter defibrillator that monitors patients at risk for SCA and provides a therapeutic shock if needed.

SUMMARY:
The Jewel IDE Study: A Clinical Evaluation of the Jewel P-WCD in Subjects at High Risk for Sudden Cardiac Arrest. ("JEWEL")

DETAILED DESCRIPTION:
Multi-center, prospective, single arm study of the Jewel Patch-Wearable Cardioverter Defibrillator (P-WCD) System in patients at high risk for Sudden Cardiac Arrest

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any gender aged ≥ 18 years.
2. Patients with either:

   1. a measured LVEF less than or equal to 40% (as assessed by techniques such as, but not limited to, cardiac angiography, echocardiography, magnetic resonance imaging, or radionuclide angiography within the last 30 days prior to enrollment) AND identified as presenting with a diagnosis of an AMI, ischemic cardiomyopathy (includes congestive heart failure: NYHA Class I - III), non- ischemic cardiomyopathy, or myocarditis;

      OR
   2. who have a temporary or long-term contraindication to receiving an ICD, who have had an ICD removed, or who refuse an ICD

      OR
   3. whose ICD implantation is delayed due to COVID-19 infection or exposure- related risks

Exclusion Criteria:

1. Member of a vulnerable patient population as defined in ISO 14155;
2. Life expectancy of less than one year, including end-stage heart failure, cancer, or other diagnosed condition;
3. Patients with an anticipated initial prescription period over 180 days (limitation only to allow timely closure of this clinical trial);
4. Patients with an advanced directive prohibiting resuscitation;
5. Existing ICD;
6. Existing unipolar pacemaker;
7. Existing FDA-cleared or FDA-approved active implantable or body worn medical device(s) that the Sponsor requires to be removed prior to the study but which cannot be removed;
8. Clinically significant valve disease, including aortic stenosis, mitral stenosis; mitral regurgitation, tricuspid regurgitation, insufficiency of the aortic or pulmonary valves, any of which is likely to require surgery in the next year;
9. A planned procedure, such as Coronary Artery Bypass Graft, within six (6) months;
10. End-stage renal disease, or chronic renal failure requiring hemodialysis;
11. Planned discharge to an institutional setting with an anticipated stay of greater than seven (7) days;
12. Having a mental, visual, physical, or auditory deficit, that could impair their ability to properly place, remove, or interact with the Jewel System;
13. Unable to understand English for the purposes of interacting with the device;
14. Unable to use a wearable defibrillator due to physical conditions (bandages preventing electrode contact, physical deformities preventing electrode contact, etc.);
15. Dextrocardia;
16. Body circumference of less than 27 inches or greater than 56 inches in the intended area of the Belt component of the Placement Accessory;
17. Participation in an investigational study of a drug, biologic, or device not currently approved for marketing;
18. Allergic to or have had a known adverse reaction to medical adhesives or hydrocolloids;
19. Active skin breakdown, erythema, or other signs of infection in the pectoral or torso regions where the Adhesive Electrode Patches are applied;
20. Females who are pregnant or breast-feeding, or planning to be pregnant in the next 12 months;
21. No US-based postal address that can be used to ship and receive study devices and supplies (a Post Office box is not an acceptable address for product shipments).
22. Patients who, in the opinion of the Investigator, are anticipated to be non-compliant with study instructions;
23. Unable to provide or have diminished capacity to provide informed consent;
24. Any condition that an Investigator believes would interfere with the intent of the study or make participation not in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, M.D., Principal Investigator — University of Mississippi Medical Center; John Hummel, M.D., Principal Investigator — Ohio State University; Roxana Mehran, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (30):
- United States (30):
  - St. Bernard's Heart and Vascular, Jonesboro, Arkansas
  - Cardiology and Medicine Clinic, P.A., Little Rock, Arkansas
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Fuqua Heart Center Piedmont Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - North Mississippi Medical Center, Tupelo, Mississippi
  - University of Mississippi Medical Center, Jackson, Missouri
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Crystal Run Healthcare - Circuit - PPDS, Middletown, New York
  - Northwell Health, New Hyde Park, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health, Winston-Salem, North Carolina
  - TriHealth Heart Institute Cardiac and Thoracic, Cincinnati, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Methodist Le Bonheur, Memphis, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Methodist Hospital, Houston, Texas
  - ACRC Trials - Hunt - PPDS, McKinney, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hummel J, Houmsse M, Tomassoni G, Nair D, Romero J, Hargrove J, Mathews K, Thakkar AB, Ullery S, Eapen ZJ, Kumar UN, Mehran R, Butler J; Jewel IDE Study Investigators. A Patch Wearable Cardioverter-Defibrillator for Patients at Risk of Sudden Cardiac Arrest. J Am Coll Cardiol. 2024 Aug 6;84(6):525-536. doi: 10.1016/j.jacc.2024.04.063. PMID 39084827

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 322
Completed | 314
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Multi-center, prospective, single arm study of the Jewel Patch-Wearable Cardioverter Defibrillator (P-WCD) System in adult subjects aged 18 years and above at high risk for Sudden Cardiac Arrest, who were not candidates for or who refused an implanted cardioverter defibrillator.
Arm/Group | Study Arm
Number analyzed (Participants) | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 302
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.0 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Inappropriate Shock Rate
Description: Inappropriate shocks no more than 2.0 inappropriate shocks per 100 patient-months.
Time Frame: Prescription Period during which each patient wore the Jewel up to 180 days.
Population: Of the 314 total patients completed, the primary analysis population was comprised of the 300 subjects who completed the study and had available device data contributing to analyzable wear time.
Measure: Number; unit: inappropriate shocks per 100 pt-months
Arm/Group | Study Arm
Number analyzed (Participants) | 300
inappropriate shocks per 100 pt-months | 0.333

2. Primary Outcome: Cutaneous Adverse Device Effects
Description: Rate of subjects experiencing clinically significant cutaneous Adverse Device Effects of < 15%
Time Frame: Prescription Period during which each patient wore the Jewel up to 180 days.
Measure: Number; unit: percentage of participants
Arm/Group | Study Arm
Number analyzed (Participants) | 314
percentage of participants | 2.23

ADVERSE EVENTS:
Time Frame: Prescription Period during which each patient wore the Jewel up to 180 days
Description: Adverse Events (AEs) defined as any untoward medical occurrence in a subject during the study that in the opinion of the investigator was at least potentially related to use of the Jewel system.
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/314
Serious Adverse Events (participants affected / at risk) | 0/314
Other Adverse Events (participants affected / at risk) | 49/314
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=314)
Skin irritation (Skin and subcutaneous tissue disorders) | 49 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT05201495/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT05201495/SAP_001.pdf